CLINICAL TRIAL: NCT05799638
Title: Medication Strategies in Heart Failure Patients Who Are Intolerable to Guideline-directed Medical Therapy
Brief Title: Strategy, Efficacy and Safety of Medication Usage in Heart Failure Patients Who Were Intolerable to GDMT
Acronym: SEMI
Status: Completed | Type: Observational
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dongying Zhang, Professor, Chongqing Medical University
Other Study IDs: SEMI-HF
Record Dates: First submitted 2023-03-12; First posted 2023-04-05 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: heart failure; myocardial fibrosis; vericiguat
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Heart Failure Patients who were tolerable to GDMT: Guideline-Directed Medication Treatment contains ACEI/ARB/ARNI, β blocker, SGLT2i and MRA. The patients in this group were tolerable to all the medications and accepted GDMT.
  Interventions: Other: Guideline-Directed Medication Treatment (GDMT)
- Heart Failure Patients who were intolerable to GDMT: The patients in this group were intolerable to one or more medication in GDMT due to hypotension, hyperkalemia or renal insufficiency.

INTERVENTIONS:
Other: Guideline-Directed Medication Treatment (GDMT) — GDMT contains ACEIs/ARBs/ARNI, β blockers, SGLT2is, MRAs. ACEI/ARB/ARNI and β blocker will gradually be titrated up to the maximum tolerable dose
  Groups: Heart Failure Patients who were tolerable to GDMT

SUMMARY:
SEMI trial is a single-center, real-world based prospective cohort study. The study enrolled acute heart failure patients admitting to the hospital and intended to accept heart failure therapy. The current guideline recommend ACEI/ARB/ARNI, β blocker, SGLT2i and MRA as the cornerstone medication of HFrEF therapy, but a part patients were intolerable to GDMT because of hypotension, hyperkalemia or renal insufficency. Vericiguat is a new medication therapy choice for the patients with heart failure with reduced ejection fraction (HFrEF), it may has less influence on blood pressure, it is unkonwn about the efficacy and safety of vericiguat in patients who were intolerable to GDMT.

DETAILED DESCRIPTION:
The study aim to provide evidence of medication strategy in heart failure patients, especially for patients who are intolerable for GDMT.

ELIGIBILITY:
Inclusion Criteria:

1. Sent to the Department of Cardiovascular disease of The First Affiliated Hospital of Chongqing Medical University for inpatient treatment.
2. Diagnosed with acute heart failure or acute exacerbation of chronic heart failure
3. Patients with typical heart failure symptoms and signs such as dyspnea, fatigue after exercise, paroxysmal nocturnal dyspnea, lower limb edema, lung auscultation rale, etc.
4. Left ventricular ejection fraction measured by echocardiogram ≤ 45% and patients had elevated level of NT-proBNP (patients<55 years, NT-proBNP>450 pg/mL; patients≥55 years and <75 years, NT-proBNP>900 pg/mL; patients ≥ 75 years, NT-proBNP>1800 pg/mL)
5. New York Heart Association functional class II to IV.

Exclusion Criteria:

1. Left ventricular ejection fraction measured by echocardiogram > 45% or diagnosed with heart failure with preserved ejection fraction.
2. Age ≤ 18 years old.
3. Allergic to anti-heart failure medications including ACEI/ARB/ARNI, beta blockers, SGLT2i, oral diuretics and vericiguat.
4. Diagnosed as other diseases with symptoms similar to heart failure such as acute exacerbation of chronic obstructive pulmonary disease, etc.
5. Dignosed with acute coronary syndrome, including unstable angina, non ST-elevation myocardial infarction and ST-elevation myocardial infarction. Received percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG) within 3 months prior to the trial start, or indication for PCI or CABG at the trial start.
6. Hepatic insufficiency classified as Child-Pugh B or C.
7. Diagnosed with restrictive cardiomyopathy.
8. Diagnosed with cardiac amyloidosis, Fabry disease or other rare cardiomyopathy.
9. Diagnosed with systematic lupus erythematosus or other autoimmune disease.
10. Diagnosed with or suspect diagnosed with active tumor.
11. Diagnosed with idiopathic pulmonary hypertension, receiving PDE-5 inhibitor or other sGC stimulators.
12. Pregnant woman.
13. Combined with severe infection at admission or combined with uncontrolled tuberculosis.
14. Diagnosed with severe and uncontrolled congenital heart disease.
15. Patients with rheumatic valvular disease who have indications for surgery but have not undergone surgical treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients enrolled in the study were recruited from a single center. The patients were admitted to hospital and diagnosed with acute heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 263 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Worsening heart failure events in 180 days | 180 days
  Risk of death, readmission due to heart failure or accepting intravenous diuretic therapy in 180 days

SECONDARY OUTCOMES:
Change in N-terminal pro-B type natriuretic peptide | 180 days
  Change in NT-proBNP level from baseline to 180 days or endpoint
Change in left ventricular ejection fraction (LVEF) | 180 days
  Change in LVEF measured by echocardiogram from baseline to 180 days or endpoint
Change in left ventricular end-diastolic diameter (LVEDD) | 180 days
  Change in LVEDD measured by echocardiogram from baseline to 180 days or endpoint
Change in left ventricular end-systolic diameter (LVESD) | 180 days
  Change in LVESD measured by echocardiogram from baseline to 180 days or endpoint
Change in left ventricular fractional shortening (LVFS) | 180 days
  Change in LVFS measured by echocardiogram from baseline to 180 days or endpoint
Change in blood pressure | 180 days
  Systolic and diastolic blood pressures were measured at admission, discharge, and up-titration to the maximum tolerated dosage
Change in blood potassium | 180 days
  Blood potassium were measured in baseline and endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Dongying Zhang, Ph.D, Study Chair — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The first affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armstrong PW, Pieske B, Anstrom KJ, Ezekowitz J, Hernandez AF, Butler J, Lam CSP, Ponikowski P, Voors AA, Jia G, McNulty SE, Patel MJ, Roessig L, Koglin J, O'Connor CM; VICTORIA Study Group. Vericiguat in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2020 May 14;382(20):1883-1893. doi: 10.1056/NEJMoa1915928. Epub 2020 Mar 28. PMID 32222134
- [Background] Armstrong PW, Roessig L, Patel MJ, Anstrom KJ, Butler J, Voors AA, Lam CSP, Ponikowski P, Temple T, Pieske B, Ezekowitz J, Hernandez AF, Koglin J, O'Connor CM. A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial of the Efficacy and Safety of the Oral Soluble Guanylate Cyclase Stimulator: The VICTORIA Trial. JACC Heart Fail. 2018 Feb;6(2):96-104. doi: 10.1016/j.jchf.2017.08.013. Epub 2017 Oct 11. PMID 29032136
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW; ACC/AHA Joint Committee Members. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2022 May 3;145(18):e895-e1032. doi: 10.1161/CIR.0000000000001063. Epub 2022 Apr 1. PMID 35363499
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Background] Mebazaa A, Davison B, Chioncel O, Cohen-Solal A, Diaz R, Filippatos G, Metra M, Ponikowski P, Sliwa K, Voors AA, Edwards C, Novosadova M, Takagi K, Damasceno A, Saidu H, Gayat E, Pang PS, Celutkiene J, Cotter G. Safety, tolerability and efficacy of up-titration of guideline-directed medical therapies for acute heart failure (STRONG-HF): a multinational, open-label, randomised, trial. Lancet. 2022 Dec 3;400(10367):1938-1952. doi: 10.1016/S0140-6736(22)02076-1. Epub 2022 Nov 7. PMID 36356631